CLINICAL TRIAL: NCT00571480
Title: Acupuncture and Low Back Pain During Pregnancy
Brief Title: Use Ear Acupuncture as Treatment for Low Back Pain During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Shu-Ming Wang, M.D., Yale University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: HIC 12291; 5R21AT001613-03 (NIH)
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2009-07

CONDITIONS: Pregnancy Related Low Back Pain
Keywords: auricular acupuncture; pregnancy related low back pain; acupuncture
MeSH Terms: interventions — Acupuncture Therapy; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 true acupuncture (Experimental): acupuncture needles are inserted into three preselected ear acupuncture points which are thought to be specific for low back pain
  Interventions: Other: acupuncture
- 2 (Sham Comparator): three acupuncture needles are inserted to three ear acupuncture points which are not specific for low back pain during pregnancy
  Interventions: Other: Sham acupuncture
- 3 (Other): standard of care
  Interventions: Other: standard of care

INTERVENTIONS:
Other: acupuncture — ear acupuncture needles will be inserted into three preselected acupuncture points which are thought to be specific for low back pain
  Other Names: retained ear acupuncture treatment
  Arms: 1 true acupuncture
Other: Sham acupuncture — ear acupuncture needles are inserted into three preselected acupuncture points which are thought not specific to low back pain
  Other Names: retained ear acupuncture treatment
  Arms: 2
Other: standard of care — participants can take acetaminophen 650 mg no more than every 6 hours and frequent rest and topical warm/cold compress
  Arms: 3

SUMMARY:
Ear acupuncture can be used as a treatment for pregnancy induced low back pain.

DETAILED DESCRIPTION:
Ear acupuncture has been used as treatment for various pain symptoms. Pregnancy related low back pain can be debilitating for pregnant women but there is lack of effective treatment. Owing to the unique circulation system between mother and fetus, prenatal care providers and gravidae are reluctant to prescribe or accept the pharmacological intervention. Thus the goal of this clinical investigation is to determine whether ear acupuncture can be used as treatment for this special clinical entity. The participants are randomized into one of the three interventions based on a computer generated randomization table. These three interventions groups are: (1) True acupuncture (2) Sham acupuncture and (3) no acupuncture. All participants are allowed to use standard of care (SOC) as a rescue treatment and the SOC consists of acetaminophen 650 mg every 6 hours no more than 4 times per day, frequent rest and topical warm/cold compress. The participants in group 1 & 2 received a total of three continuous retained ear acupuncture needles at three sites ipsilateral to the dominant hand in preselected ear acupuncture points for one week then after day 7. All participants are followed/observed for a total 2 weeks after the initiation of the study.

ELIGIBILITY:
Inclusion Criteria:

* English speaking, healthy pregnant women in at least 25 weeks of gestational age who suffered from low back pain related to pregnancy.
* No obstetric complications during pregnancy or neurological complications that require immediate medical/surgical intervention.

Exclusion Criteria:

* Non-English speaking
* Mentally challenged
* State of pregnancy less than 25 weeks but suffer from pregnancy related low back pain
* Pregnant women without low back pain
* The pregnancy is complicated by obstetrical problems, or low back pain requiring immediate surgical/medical intervention.

Ages: 13 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 159 (Actual)
Dates: Start 2005-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
severity pain | two weeks

SECONDARY OUTCOMES:
daily disability index | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Ming Wang, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States